CLINICAL TRIAL: NCT01012726
Title: FIST-MC-09 Study About the Effect of Doxycycline and Acetylcystein in the Treatment of CD-associated Fistulae
Brief Title: Study About the Effect of Doxycycline and Acetylcystein in the Treatment of CD-associated Fistulae
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough patients enrolled
Sponsor: Gerhard Rogler (Other)
Responsible Party: Sponsor-Investigator, Gerhard Rogler, Prof. Dr. Dr. Gerhard Rogler, University of Zurich
Organization: University of Zurich (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIST-MC-09
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Colonoscopy

INTERVENTIONS:
Procedure: Colonoscopy — During the colonoscopy, we instill Acetylcystein and Doxycyline into the fistula.

SUMMARY:
The investigators will study whether local instillation of Doxycycline and Acetylcystein results in fistula closure in CD patients.

ELIGIBILITY:
Inclusion criteria:

* fistulizing CD
* CD < 6 months
* at least one insufficient fistula closure try

Exclusion criteria:

* CDAI > 200
* Abscesses
* CRP > 100

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Fistula closure | 01.08.2009 - 31.07.2012

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland